CLINICAL TRIAL: NCT06138301
Title: Digital Interventions for Social isOLation In youThs And theIR familiEs
Brief Title: Telepsychiatry for Social Isolation in Youths
Acronym: SOLITAIRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Collaborators: IRCCS Eugenio Medea (Other); University of Milan (Other); Istituto di Neuroscienze Consiglio Nazionale delle Ricerche (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4202CESC; PNRR-MAD-2022-12376834 (Other Grant/Funding Number: European Union - Next Generation EU - NRRP M6C2)
Record Dates: First submitted 2023-09-04; First posted 2023-11-18 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Social Isolation; Psychosocial Problem
Keywords: Social Isolation; Telepsychiatry; Digital health; Cognitive remediation; CBT; Psychotherapy; Loneliness
MeSH Terms: conditions — Social Isolation | interventions — Cognitive Behavioral Therapy; Cognitive Remediation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patients with SI treated with CBT+CR
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT); Behavioral: Cognitive Remediation (CR)
- Control group (Active Comparator): Patients with SI treated with CBT
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) — CBT is a psychotherapeutic intervention that focuses on challenging and changing cognitive distortions (such as thoughts, beliefs, and attitudes) and their associated behaviours to improve emotional regulation and develop personal coping strategies that target solving current problems. In this study, patients with SI will undergo 8 sessions of CBT (45 min, once a week), remotely. Techniques and strategies of the intervention will be based on a short telepsychotherapy protocol previously published by our group (Biagianti et. al., 2021). Instead, the content of each session will be adapted to the psychopathology associated with social isolation and the age of the subject. The psychotherapeutic sessions of the patients will be audio-recorded in order to conduct retrospective analyzes of the patient's speech.
Behavioral: Cognitive Remediation (CR) — The cognitive training will consist of 10 hours (30 minutes/session) of computer-based exercises focusing on working memory, attention, executive functions and social cognition, which will be performed online using BrainHQ software. This software allows for the customization of the training based on the specific characteristics of each subject. For example, it allows automatic adjustment of the difficulty of the exercises, trial by trial and session by session, in order to guarantee an adequate level of attention and motivation for the entire duration of the training and therefore favor optimal learning rates.
  Arms: Experimental group

SUMMARY:
This clinical trial aims to implement multimodal digital interventions for adolescents and young adults with social isolation (SI) and their family members. Furthermore, the neurobiological basis of SI will be explored by analyzing blood neuroinflammation biomarkers in socially isolated participants.

The main questions that this project aims to answer are:

* What is the general feasibility and applicability of the proposed digital interventions?
* What is the effect of the proposed digital interventions on the SI-related clinical symptoms and the cognitive and global functioning of participants with SI?

Participants will be asked to undergo:

* A detailed clinical and neuropsychological evaluation (pre-post treatment)
* A blood sample (pre-post treatment)
* A telepsychiatry intervention (cognitive behavioural therapy (CBT) and/or cognitive remediation (CR) for SI participants and psychoeducation (PE) for family members)

The researchers will compare SI participants treated with CBT+CR (experimental group) with SI patients treated only with CBT (control group) to see if the combined intervention of the experimental group leads to more durable and generalizable effects.

The same PE intervention will be offered to the family members of all recruited SI participants.

DETAILED DESCRIPTION:
SI is a condition that can lead to complete withdrawal from society, especially concerning the most fragile subgroups, such as youth and elderly populations. It is often a core (often prodromal) symptom of severe psychiatric disorders such as Hikikomori syndrome, social anxiety disorder, psychosis, depression, post-traumatic disorders stress disorder, obsessive-compulsive disorder, mood dysregulation, and autism spectrum disorders. If left untreated, SI can escalate into complete withdrawal from society. Therefore, early interventions for the treatment of SI could lead to a more favourable outcome for young patients. However, due to the social interaction barrier inherent to the condition, current treatments alone are problematic and only partially effective in treating SI. SOLITAIRE aims to implement a multi-component digital psychiatric intervention to help adolescents and young adults with SI based on CBT and/or CR for socially isolated participants and PE for their family members. All interventions will be delivered remotely, thus overcoming most of the barriers and limitations of standard face-to-face clinical interventions. In particular, a randomized controlled trial (RCT) will be conducted on participants with SI to test the feasibility and acceptability of the interventions and to evaluate the difference in efficacy between CBT+CR (experimental group) and CBT alone (control group). The CBT sessions will be audio-recorded. The recordings will then be analyzed using machine learning algorithms to build an automatic system for the evaluation of SI-related depressive symptoms starting from the voice. The digital interventions will last about 2-3 months. The investigators hypothesized that participants in the experimental group would show more durable and generalizable cognitive and behavioural improvements due to the neuroplasticity processes associated with CR. Furthermore, plasma samples of the socially isolated participants will be collected before and after the interventions and biochemically analyzed to explore the neurobiological basis of SI and treatment-related biomarkers.

Family members will be invited to undergo video calls with a psychotherapist (8 sessions, ≈1 hour/week) in which cognitive-behavioural and PE techniques will be combined to provide them with knowledge about the clinical aspects and treatments of SI. The content of the sessions will be adapted to the age and specific psychopathological profile of the socially isolated relatives.

Participants with SI can be included in the study even if their family members choose not to participate.

ELIGIBILITY:
Inclusion Criteria:

Patients with SI:

* age11-17 years (adolescents) 18-45 years (adults)
* moderate-to-high levels of SI as detected by clinical evaluation and confirmed by the HQ-25 score
* stable pharmacotherapy and symptomatology in the last 3 months
* not being in psychotherapy or being willing to interrupt it during the study
* have an internet connection

Caregivers:

* Age ≤ 80
* no history of psychotic spectrum disorders
* have a first-degree relative with moderate-to-severe SI
* have an internet connection

Exclusion Criteria:

All participants:

* primary medical conditions or vision/hearing deficits that interfere with the ability to participate in the project
* suicidal Ideation
* IQ < 70

Ages: 11 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Change in SI-related symptoms in socially isolated participants, as assessed by the Hikikomori Questionnaire (HQ-25); [score range 0-100; higher scores mean worse outcome]. | up to 4 months
  Response to treatment is defined as a post-pre treatment reduction ≥ 25% in the HQ-25 score
Feasibility and acceptability of the digital interventions | up to 4 months
  I) The completion rate of the baseline and follow-up assessments ii) the completion rate of the entire study (completers vs drop-outs).
Usability of the digital interventions | up to 4 months
  Scores obtained on a 7pt Likert scale created ad hoc

SECONDARY OUTCOMES:
Change in the clinical and cognitive profile of socially isolated participants. | up to 4 months
  Post-pre treatment mean change in the score of questionnaires/tests measuring depression, anxiety, alexithymia, behaviour, loneliness, social interaction, impulsivity, temperament and character, close relationships, quality of life, general health, functioning, psychological needs and parental bonding as well as attention, memory, executive functions and linguistic comprehension.
  Depending on the questionnaire/test taken into consideration, higher scores can mean either a better or worse outcome. Therefore, the scores of the various questionnaires/tests will be standardized (e.g., z-transformed) to allow for comparisons.
Change in psychological burden and well-being of family members as assessed by self-report questionnaires. | up to 4 months
  Post-pre treatment mean change in the questionnaire scores. Depending on the questionnaire/test taken into consideration, higher scores can mean either a better or worse outcome. Therefore, the scores of the various questionnaires/tests will be standardized (e.g., z-transformed) to allow for comparisons.
Change of SI-related depressive symptoms measured via speech analysis | up to 4 months
  CBT sessions will be audio recorded. The recordings will then be analyzed using machine learning algorithms to build an automatic system for the evaluation of SI-related depressive symptoms starting from the voice. The scores produced by the automatic algorithm will be compared during the 8 weeks of intervention. Since these are exploratory analyses, these scores will be defined during the research itself (there are no widely accepted standard methodologies for this type of innovative analysis).
Identification of plasmatic biomarkers related to social isolation pathology and treatment | up to 4 months
  Blood samples of the participants will be collected before (T0) and at the end of (T1) the treatments. Blood serum will be analyzed through a Luminex200 multiplex immunoassay to quantify the levels of selected proteins. These will include markers previously reported to be altered in psychiatric conditions, such as BDNF, EGF, RANTES, MMP-9, IL-1, IL-6, TGFalpha.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Mirella Ruggeri, PhD, Principal Investigator — Section of Psychiatry, University of Verona
Locations (2):
- Italy (2):
  - Unità per le Disabilità gravi dell'età Evolutiva e Giovane Adulta, IRCCS Eugenio Medea, Polo scientifico Puglia, Brindisi
  - UOC Psichiatria B, Azienda Ospedaliera Universitaria Integrata, Verona

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie behavioural results, after deidentification(text, tables, figures, and appendices)
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Immediately following publication.No end date.
Access Criteria: Proposals should be directed to marcella.bellani@univr.it. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Bhatti AB, Haq AU. The Pathophysiology of Perceived Social Isolation: Effects on Health and Mortality. Cureus. 2017 Jan 24;9(1):e994. doi: 10.7759/cureus.994. PMID 28382237
- [Background] Biagianti B, Zito S, Fornoni C, Ginex V, Bellani M, Bressi C, Brambilla P. Developing a Brief Tele-Psychotherapy Model for COVID-19 Patients and Their Family Members. Front Psychol. 2021 Dec 2;12:784685. doi: 10.3389/fpsyg.2021.784685. eCollection 2021. PMID 34925187
- [Background] Cacioppo S, Capitanio JP, Cacioppo JT. Toward a neurology of loneliness. Psychol Bull. 2014 Nov;140(6):1464-504. doi: 10.1037/a0037618. Epub 2014 Sep 15. PMID 25222636
- [Background] De France K, Hancock GR, Stack DM, Serbin LA, Hollenstein T. The mental health implications of COVID-19 for adolescents: Follow-up of a four-wave longitudinal study during the pandemic. Am Psychol. 2022 Jan;77(1):85-99. doi: 10.1037/amp0000838. Epub 2021 May 24. PMID 34110880
- [Background] Domenici E, Wille DR, Tozzi F, Prokopenko I, Miller S, McKeown A, Brittain C, Rujescu D, Giegling I, Turck CW, Holsboer F, Bullmore ET, Middleton L, Merlo-Pich E, Alexander RC, Muglia P. Plasma protein biomarkers for depression and schizophrenia by multi analyte profiling of case-control collections. PLoS One. 2010 Feb 11;5(2):e9166. doi: 10.1371/journal.pone.0009166. PMID 20161799
- [Background] Faurholt-Jepsen M, Busk J, Frost M, Vinberg M, Christensen EM, Winther O, Bardram JE, Kessing LV. Voice analysis as an objective state marker in bipolar disorder. Transl Psychiatry. 2016 Jul 19;6(7):e856. doi: 10.1038/tp.2016.123. PMID 27434490
- [Background] Garcia-Gutierrez MS, Navarrete F, Sala F, Gasparyan A, Austrich-Olivares A, Manzanares J. Biomarkers in Psychiatry: Concept, Definition, Types and Relevance to the Clinical Reality. Front Psychiatry. 2020 May 15;11:432. doi: 10.3389/fpsyt.2020.00432. eCollection 2020. PMID 32499729
- [Background] Gershkovich M, Herbert JD, Forman EM, Schumacher LM, Fischer LE. Internet-Delivered Acceptance-Based Cognitive-Behavioral Intervention for Social Anxiety Disorder With and Without Therapist Support: A Randomized Trial. Behav Modif. 2017 Sep;41(5):583-608. doi: 10.1177/0145445517694457. Epub 2017 Mar 8. PMID 28776431
- [Background] Low DM, Bentley KH, Ghosh SS. Automated assessment of psychiatric disorders using speech: A systematic review. Laryngoscope Investig Otolaryngol. 2020 Jan 31;5(1):96-116. doi: 10.1002/lio2.354. eCollection 2020 Feb. PMID 32128436
- [Background] McEvoy PM. Effectiveness of cognitive behavioural group therapy for social phobia in a community clinic: a benchmarking study. Behav Res Ther. 2007 Dec;45(12):3030-40. doi: 10.1016/j.brat.2007.08.002. Epub 2007 Aug 8. PMID 17826734
- [Background] Merikangas KR, He JP, Burstein M, Swendsen J, Avenevoli S, Case B, Georgiades K, Heaton L, Swanson S, Olfson M. Service utilization for lifetime mental disorders in U.S. adolescents: results of the National Comorbidity Survey-Adolescent Supplement (NCS-A). J Am Acad Child Adolesc Psychiatry. 2011 Jan;50(1):32-45. doi: 10.1016/j.jaac.2010.10.006. Epub 2010 Dec 3. PMID 21156268
- [Background] Nagata T, Yamada H, Teo AR, Yoshimura C, Nakajima T, van Vliet I. Comorbid social withdrawal (hikikomori) in outpatients with social anxiety disorder: clinical characteristics and treatment response in a case series. Int J Soc Psychiatry. 2013 Feb;59(1):73-8. doi: 10.1177/0020764011423184. Epub 2011 Oct 13. PMID 21997765
- [Background] Nordh M, Vigerland S, Ost LG, Ljotsson B, Mataix-Cols D, Serlachius E, Hogstrom J. Therapist-guided internet-delivered cognitive-behavioural therapy supplemented with group exposure sessions for adolescents with social anxiety disorder: a feasibility trial. BMJ Open. 2017 Dec 14;7(12):e018345. doi: 10.1136/bmjopen-2017-018345. PMID 29247101
- [Background] Kim EJ, Bahk YC, Oh H, Lee WH, Lee JS, Choi KH. Current Status of Cognitive Remediation for Psychiatric Disorders: A Review. Front Psychiatry. 2018 Oct 1;9:461. doi: 10.3389/fpsyt.2018.00461. eCollection 2018. PMID 30337888
- [Background] Ramdhani, N., Widjaja, J. D., & Rahmawati, N. (2015). Internet supported cognitive behavior therapy to help students with shy-socially isolated problems. Procedia-Social and Behavioral Sciences, 165, 179-188.
- [Background] Rohr S, Wittmann F, Engel C, Enzenbach C, Witte AV, Villringer A, Loffler M, Riedel-Heller SG. Social factors and the prevalence of social isolation in a population-based adult cohort. Soc Psychiatry Psychiatr Epidemiol. 2022 Oct;57(10):1959-1968. doi: 10.1007/s00127-021-02174-x. Epub 2021 Sep 17. PMID 34533607
- [Background] Sarkhel S, Singh OP, Arora M. Clinical Practice Guidelines for Psychoeducation in Psychiatric Disorders General Principles of Psychoeducation. Indian J Psychiatry. 2020 Jan;62(Suppl 2):S319-S323. doi: 10.4103/psychiatry.IndianJPsychiatry_780_19. Epub 2020 Jan 17. No abstract available. PMID 32055073
- [Background] Strawbridge R, Young AH, Cleare AJ. Biomarkers for depression: recent insights, current challenges and future prospects. Neuropsychiatr Dis Treat. 2017 May 10;13:1245-1262. doi: 10.2147/NDT.S114542. eCollection 2017. PMID 28546750
- [Background] Taylor HO, Taylor RJ, Nguyen AW, Chatters L. Social Isolation, Depression, and Psychological Distress Among Older Adults. J Aging Health. 2018 Feb;30(2):229-246. doi: 10.1177/0898264316673511. Epub 2016 Oct 17. PMID 28553785
- [Background] Teo AR. Social isolation associated with depression: a case report of hikikomori. Int J Soc Psychiatry. 2013 Jun;59(4):339-41. doi: 10.1177/0020764012437128. Epub 2012 Mar 8. PMID 22408115
- [Background] Wang J, Zhang L, Liu T, Pan W, Hu B, Zhu T. Acoustic differences between healthy and depressed people: a cross-situation study. BMC Psychiatry. 2019 Oct 15;19(1):300. doi: 10.1186/s12888-019-2300-7. PMID 31615470
- [Background] Zovetti N, Rossetti MG, Perlini C, Brambilla P, Bellani M. Neuroimaging studies exploring the neural basis of social isolation. Epidemiol Psychiatr Sci. 2021 Apr 6;30:e29. doi: 10.1017/S2045796021000135. PMID 33820592